CLINICAL TRIAL: NCT01727362
Title: Evaluation of Effectiveness of Acupuncture on Quality of Life in Patients With Breast Cancer Receiving Chemotherapy- A Pragmatic Randomized Trial
Brief Title: Evaluation of Effectiveness of Acupuncture on Quality of Life in Patients With Breast Cancer Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Mammazentrum Hamburg am Krankenhaus Jerusalem, Germany (Unknown); Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Professor, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACU in breast cancer
Record Dates: First submitted 2012-11-07; First posted 2012-11-16 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Acupuncture; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care + acupuncture (Active Comparator)
  Interventions: Other: Usual care + acupuncture
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care + acupuncture — Patients of this group receive a semi-standardized acupuncture treatment over 6 month in addition to usual care
  Arms: Usual care + acupuncture
Other: Usual care — Patients of this group receive usual care only
  Arms: Usual care

SUMMARY:
The aim of this trial is to investigate the effectiveness of acupuncture on quality of life in patients with breast cancer receiving chemotherapy compared to routine care.

DETAILED DESCRIPTION:
At the Mammazentrum Hamburg, Germany, patients with breast cancer receiving chemotherapy have the opportunity to get acupuncture in addition to conventional therapy to maintain quality of life and to reduce the side effects of the chemotherapy such as gastrointestinal disorders. In this randomized trial we aim to investigate the effectiveness of additional acupuncture compared to routine care in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed breast cancer (invasive, intraductal, hormone-sensitive and not hormone-sensitive, only locoregional metastases)
* current chemotherapy at Mammazentrum Hamburg with regimen FEC/DOC or EC/DOC
* willingness to receive acupuncture within the next 6 month if randomized in acupuncture group
* willingness to refrain from acupuncture within the next 6 month if randomized in control group
* informed consent

Exclusion Criteria:

* distant metastases
* blood coagulation disorder and/or current use of anticoagulants
* serious acute or chronic mental or physical disorders
* clinically relevant cardiac arrhythmia symptoms
* insufficient German language ability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | 6 month

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | 3 month

OTHER OUTCOMES:
Subscales of the Functional Assessment of Cancer Therapy - General (FACT-G): physical well-being, social/family well-being, emotional well-being, functional well-being | 3 month
Subscales of the Functional Assessment of Cancer Therapy - General (FACT-G): physical well-being, social/family well-being, emotional well-being, functional well-being | 6 month
Subscale for Breast Cancer of the Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | 3 month
Subscale for Breast Cancer of the Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | 6 month
Pain, quality of sleep, and nausea (single items of the FACT-B) | 3 month
Pain, quality of sleep, and nausea (single items of the FACT-B) | 6 month
Functional Assessment of Chronic Illness Therapy-Fatigue | 3 month
Functional Assessment of Chronic Illness Therapy-Fatigue | 6 month
FACT/GOG-NTX, polyneuropathy symptoms | 3 month
FACT/GOG-NTX, polyneuropathy symptoms | 6 month
Quality of Life (SF-12 Health Survey) | 3 month
Quality of Life (SF-12 Health Survey) | 6 month
Survival without relapse | 6 month
Survival | 6 month
Adverse effects and Interactions | 3 month
Adverse effects and Interactions | 6 month
Satisfaction and patient-reported effectiveness | 3 month
  This will only be assessed in the acupuncture arm
Satisfaction and patient-reported effectiveness | 6 month
  This will only be assessed in the acupuncture arm
Goal Attainment Scale | 3 month
  This will only be assessed in the acupuncture arm
Goal Attainment Scale | 6 month
  This will only be assessed in the acupuncture arm
Laboratory parameters (hemoglobin, leukocytes, blood plates, liver values, kidney values) | 3 month
Laboratory parameters (hemoglobin, leukocytes, blood plates, liver values, kidney values) | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Martin Carstensen, Prof. MD, Principal Investigator — Mammazentrum am Krankenhaus Jerusalem, Hamburg, Germany
Locations (1):
- Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg, Germany

REFERENCES:
- [Derived] Stockigt DMB, Kirschbaum B, Carstensen DMM, Witt DMCM, Brinkhaus DMB. Prophylactic Acupuncture Treatment During Chemotherapy in Patients With Breast Cancer: Results of a Qualitative Study Nested in a Randomized Pragmatic Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211058207. doi: 10.1177/15347354211058207. PMID 34814766
- [Derived] Brinkhaus B, Kirschbaum B, Stockigt B, Binting S, Roll S, Carstensen M, Witt CM. Prophylactic acupuncture treatment during chemotherapy with breast cancer: a randomized pragmatic trial with a retrospective nested qualitative study. Breast Cancer Res Treat. 2019 Dec;178(3):617-628. doi: 10.1007/s10549-019-05431-5. Epub 2019 Sep 13. PMID 31520284